CLINICAL TRIAL: NCT06315842
Title: Levels of Diagnostic and Therapeutic Intervention in Hospitalized Patients. Cluster-Randomized and Stepped-Wedge Clinical Trial
Brief Title: Levels of Diagnostic and Therapeutic Intervention in Hospitalized Patients
Acronym: NIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: CSAPG-44
Record Dates: First submitted 2024-03-05; First posted 2024-03-18 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Acute Disease
Keywords: Patient Care Planning; Decision Making; Advance Care Planning
MeSH Terms: conditions — Acute Disease | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Intervention Model Description: The participating physicians will be grouped into 4 clusters (5 physicians each). Each cluster will progressively (every 3 months) incorporate the use of a level of diagnostic and therapeutic intensity tool into their usual clinical practice.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levels of Diagnostic and Therapeutic Intervention tool (Experimental): Medical doctors assigned to this group will incorporate a Levels of Diagnostic and Therapeutic Intervention tool into their clinical practice
  Interventions: Other: Levels of Diagnostic and Therapeutic Intervention tool by Fontecha and col.
- Usual clinical practice (Active Comparator): Medical doctors assigned to this group will continue their clinical practice as usual
  Interventions: Other: Usual clinical practice

INTERVENTIONS:
Other: Levels of Diagnostic and Therapeutic Intervention tool by Fontecha and col. — During the intervention periods, participating physicians will integrate into their usual clinical practice a tool for adjusting diagnostic and therapeutic intensity designed by Fontecha-Gómez and colleagues. The tool for adjusting the level of diagnostic and therapeutic intensity classifies patients' profiles into 5 groups based on the recommended level of adjustment.
  Arms: Levels of Diagnostic and Therapeutic Intervention tool
Other: Usual clinical practice — The participating physicians will carry out the standard clinical practice currently performed in the study centers. This means that during this period, the diagnostic and therapeutic adjustment tool or any similar tool will not be introduced into routine clinical practice.
  Arms: Usual clinical practice

SUMMARY:
The objective of this clinical trial is to investigate the impact of implementing a tool for adjusting the level of diagnostic and therapeutic intensity in the clinical practice of physicians attending hospitalized patients.

The goal of this clinical trial is to investigate the impact of a tool for adjusting diagnostic and therapeutic intensity in hospitalized patients. The main question it aims to answer is: Is there a difference in patient mortality when using the aforementioned tool? The participating physicians will be grouped into 4 groups (5 physicians each). Each group will progressively (every 3 months) incorporate the use of the aforementioned tool into their usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Physician belonging to the non-surgical medical area.
* Routine clinical activity on a hospital ward caring for hospitalized patients.

Exclusion Criteria:

* Physician belonging to the Oncology-Hematology/Palliative Care Hospitalization Unit.
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
In-hospital Patient Mortality at 90 days from hospital discharge | 90 days from hospital discharge
  Percentage of patients who die during hospitalization until 90 days from hospital discharge.

SECONDARY OUTCOMES:
In-hospital Patient Mortality at 6 months from hospital discharge | 6 months from hospital discharge
  Percentage of patients who die during hospitalization until 6 months from hospital discharge.
In-hospital Patient Mortality at 1 year from hospital discharge | 1 year from hospital discharge
  Percentage of patients who die during hospitalization until 1 year from hospital discharge.
Delirium Incidence | hospital discharge, assessed up to day 90
  Percentage of patients with delirium occurrence during hospital admission (delirium already present at the time of admission will not be considered). Delirium will be evaluated through Confusion Assessment Method (CAM)
Pressure Ulcer Incidence | hospital discharge, assessed up to day 90
  Percentage of patients with pressure ulcer occurrence during hospital admission (pressure ulcers already present at the time of admission will not be considered).
Hospital stay | hospital discharge, assessed up to day 90
  Hospital stay in days
Hospital readmission for any reason | 30 days from hospital discharge
  Percentage of patients readmitted for any reason within 30 days of hospital discharge.
Hospital readmission for same reason | 30 days from hospital discharge
  Percentage of patients readmitted for the same reason within 30 days of hospital discharge.
Patients admitted to the Intensive Care Unit (ICU) | hospital discharge, assessed up to day 90
  Percentage of patients admitted to the ICU during hospitalization
Calls to the "on-call doctor" | hospital discharge, assessed up to day 90
  Number of calls to the "on-call doctor" during hospital admission
Healthcare expenditure | through study completion, an average of 1.5 years
  Descriptive analysis of healthcare expenditure associated with each intervention, using the billing data from the center.
Mortality at ICU | hospital discharge, assessed up to day 90
  Percentage of patients admitted to the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Helena Camell, Principal Investigator — CSAPG; César Gálvez, Study Director — CSAPG
Locations (1):
- Consorci Sanitari Alt Penedes i Garraf, Vilafranca del Penedès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research proposels and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.

REFERENCES:
- [Background] Fontecha-Gomez BJ, Amblas-Novellas J, Betancor-Santana E, Rexach-Cano L, Ugarte MI, Lopez-Perez A, Planas K, Gutierrez Jimenez N, Casas Floriano R, Garcia-Fortea C, Serrano Bermudez G, Rotllan-Terradellas M, Fernandez-Ponce D. [Regional protocol for adjusting the therapeutic intensity. Southern Metropolitan Area of Barcelona]. Rev Esp Geriatr Gerontol. 2018 Jul-Aug;53(4):217-222. doi: 10.1016/j.regg.2018.01.003. Epub 2018 Feb 21. Spanish. PMID 29475629